CLINICAL TRIAL: NCT06842108
Title: Relationship Between Hemodynamic Changes and Cardiopulmonary Fitness in Type 2 Diabetes Mellitus Patients
Acronym: diabetes
Status: Recruiting | Type: Observational
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Seyyada Tahniat Ali, physiotherapist, Bahria University
Other Study IDs: 122/24
Record Dates: First submitted 2025-02-13; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus Type 2 (T2DM)
Keywords: Diabetes Mellitus; Hemodynamic changes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Controlled type 2 Diabetes Mellitus patients.: The data will be collected after taking consent from patients who will be undergoing ETT.
  Interventions: Other: Exercise tolerance test

INTERVENTIONS:
Other: Exercise tolerance test — • The ETT will be performed using Bruce protocol. The Bruce protocol is a standardized treadmill exercise test used in Exercise Tolerance Testing (ETT) to evaluate cardiovascular fitness and diagnose heart conditions. This protocol is divided into seven stages, each stage duration is 3 minutes and date will be recorded at the end of the each stage. The recorded data will include heart Rate, Rate pressure product (∆RPP), HRR1 and Blood Pressure.
  STEP 1:
  Patient Preparation
  STEP 2:
  Consent and history:
  STEP 3:
  Start of ETT:
  • Graded Exercise
  STEP 4:
  Parameters Recorded During ETT:
  * Heart Rate: Monitoring heart rate response to exercise stress.
  * Exercise induced changes in heart rate (∆HR) along with change in rate pressure product (∆RPP) due to excercise intensity.
  STEP 5:
  Cardiopulmonary Fitness Assessment VO2 Max

SUMMARY:
Diabetes mellitus being metabolic disorder, chronic in nature, is characterized by high levels of glucose in our blood, which often lead to organ dysfunction. Approximately 10.5 % of adult (20-79 years) have diabetes according to international Diabetes federation. Cardiorespiratory fitness (CRF) is the capability of our cardiopulmonary system to make oxygen available to our skeletal muscles during physical activities for prolonged time, and is known to be decreased with diabetes. Hemodynamic parameters are correlated with various cardiovascular disorders but little evidence of hemodynamic changes in diabetes patients is present and more studies must be done. This study aims to establish the link between hemodynamic changes and cardiopulmonary fitness in T2DM patients, which could inform clinical practices and interventions to improve management, reduce cardiovascular risks, and enhance the quality of life for these patients.

DETAILED DESCRIPTION:
Diabetes mellitus being metabolic disorder, chronic in nature, is characterized by high levels of glucose in our blood, which often lead to organ dysfunction.[1] Diabetes statistics highlight the increasing worldwide impact on individuals, families and nations. Approximately 10.5 % of adult (20-79 years) have diabetes according to international Diabetes federation. [2] Cardiorespiratory fitness (CRF) is the capability of our cardiopulmonary system to make oxygen available to our skeletal muscles during physical activities for prolonged time. [3] Diabetes and cardiorespiratory fitness are inter related. According to a 2023 studies on Cardiorespiratory fitness in individuals with T2DM, it was found that T2DM was associated with decreased cardiorespiratory fitness.

Hemodynamic characteristics have been linked to diseases like stroke,, hypertension, and vascular stenosis. Only a few modest studies have investigated the relationship between hemodynamics and diabetes mellitus (DM). The evidence for a link between hemodynamic alterations and CRF in type 2 diabetic individuals needs to be demonstrated. The study aimed to identify the relationship between hemodynamic changes and CRF in type 2 diabetic patients; the findings will help us form inform clinical practices and intervention strategies, ultimately leading to better T2DM management, lowering the risk of cardiovascular complications, and improving T2DM patients' quality of life and longevity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who agreed to sign the informed consent form.
* Subject with an age group 30-50yrs.
* Female and male.
* Controlled type 2 Diabetes Mellitus patients.

Exclusion Criteria:

* Patient performing any exercise.
* cardiovascular diseases.
* Patients with Cerebrovascular diseases.
* Patients with Peripheral artery diseases.
* Patients with pulmonary dysfunction.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Type 2 diabetes mellitus patients
Sampling Method: Non-Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
hemodynamic changes | Immediately after performing test
  it will be assessed through ΔHeart Rate and HRR1
Cardiorespiratory fitness | immediately after performing test
  it will be measured from VO2 max.

CONTACTS AND LOCATIONS:
Locations (1):
- bahria university Health sciences campus karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Mhanna SB, Batrakoulis A, Wan Ghazali WS, Mohamed M, Aldayel A, Alhussain MH, Afolabi HA, Wada Y, Gulu M, Elkholi S, Abubakar BD, Rojas-Valverde D. Effects of combined aerobic and resistance training on glycemic control, blood pressure, inflammation, cardiorespiratory fitness and quality of life in patients with type 2 diabetes and overweight/obesity: a systematic review and meta-analysis. PeerJ. 2024 Jun 14;12:e17525. doi: 10.7717/peerj.17525. eCollection 2024. PMID 38887616